CLINICAL TRIAL: NCT03655964
Title: Olmesartan Versus Nebivolol in Management of Hypertension in Acute Ischemic Stroke
Brief Title: Effect of Olmesartan and Nebivolol on Ambulatory Blood Pressure and Arterial Stiffness in Acute Stage of Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Vaios Vasileios, Principal Investigator, Division of Nephrology and Hypertension, 1st Department of Medicine, AHEPA University Hospital, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3418
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — olmesartan; Nebivolol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Olmesartan (Experimental): 20 patients randomly allocated to single-blind antihypertensive therapy with olmesartan (20 mg/day)
  Interventions: Drug: Olmesartan
- Nebivolol (Experimental): 20 patients randomly allocated to single-blind antihypertensive therapy with nebivolol (5 mg/day)
  Interventions: Drug: Nebivolol
- No antihypertensive treatment (Experimental): 20 patients randomly allocated to receive no antihypertensive therapy during the acute stage of ischemic stroke
  Interventions: Other: No antihypertensive treatment

INTERVENTIONS:
Drug: Olmesartan — At Day 4 of stroke onset, patients with clinic BP >160/100 mmHg will receive olmesartan 20 mg once daily until Day 7 of stroke onset
  Other Names: No other intervention
  Arms: Olmesartan
Drug: Nebivolol — At Day 4 of stroke onset, patients with clinic BP >160/100 mmHg will receive nebivolol 5mg once daily until Day 7 of stroke onset
  Other Names: No other intervention
  Arms: Nebivolol
Other: No antihypertensive treatment — Patients will be left without treatment
  Other Names: No other intervention
  Arms: No antihypertensive treatment

SUMMARY:
Single-blind, randomized, active-treatment controlled clinical study evaluating the effect of omesartan and nebivolol versus no treatment on 24-hour brachial and central aortic blood pressure in hypertensive patients with acute ischemic stroke

DETAILED DESCRIPTION:
A total of 60 patients with hypertension and acute ischemic stroke (clinic BP >160/100 mmHg and <220/120 mmHg at day 3 of stroke onset) will be randomly allocated to therapy with olmesartan (20 mg/day) or nebivolol (5 mg/day) or no treatment between the 3rd to 7th day of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a first diagnosis of an acute ischemic stroke (permanent or transient)
2. BP levels >160/100mmHg at start of the third day of hospitalization
3. BP levels >160/100mmHg and <220/120mmHg at start of the fourth day of hospitalization

Exclusion Criteria:

1. Patients with confirmed hemorrhagic stroke with computer tomography at hospital admission.
2. Patients with chronic atrial fibrillation or other cardiac arrhythmia.
3. Patients with BP levels >220/120 mmHg during the hospitalization or patients with other hypertensive emergency situation (i.e. acute myocardial ischemia, aortic dissection, acute pulmonary edema, acute renal failure, hypertensive encephalopathy) which demands fast BP reduction with the use of intravenous antihypertensive drugs, according to current guidelines {Jauch, 2013 340 /id}.
4. Patients with specific indication for treatment with blockers of the renin-angiotensin-aldosterone system (RAAS) other than hypertension (i.e., congestive heart failure, acute myocardial ischemia).
5. Patients with specific indication for treatment with β-blockers other than hypertension (i.e., heart failure, tachyarrhythmia or angina pectoris).
6. Patients with specific contra-indications for RAAS blockers (hyperkalemia, history of angioedema) and patients with a history of allergic reaction or severe hypotension after olmesartan treatment.
7. Patients with specific contra-indications for β-blockers (heart rate <60/min without a treatment with bradyarrhythmic drugs), chronic obstructive pulmonary disease or asthma and patients with history of allergic reaction after nebivolol treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Between-group difference in change of 24-hour brachial BP | Day 3 until Day 7 of stroke onset
  24-hour ambulatory BP monitoring with the Mobil-O-Graph device (IEM, Germany) at baseline (Day 3 of stroke onset) and study-end (Day 7 of stroke onset)

SECONDARY OUTCOMES:
Between-group difference in change of 24-hour pulse wave velocity | Day 3 until Day 7 of stroke onset
  24-hour ambulatory BP monitoring with the Mobil-O-Graph device (IEM, Germany) at baseline (Day 3 of stroke onset) and study-end (Day 7 on stroke onset)
Between-group difference in change of 24-hour augmentation index | Day 3 until Day 7 of stroke onset
  24-hour ambulatory BP monitoring with the Mobil-O-Graph device (IEM, Germany) at baseline (Day 3 of stroke onset) and study-end (Day 7 on stroke onset)
Between-group difference in 24-hour central aortic BP | Day 3 until Day 7 of stroke onset
  24-hour ambulatory BP monitoring with the Mobil-O-Graph device (IEM, Germany) at baseline (Day 3 of stroke onset) and study-end (Day 7 on stroke onset)

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Georgianou, MD, Principal Investigator — School of Medicine, Aristotle University of Thessaloniki
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lobanova I, Qureshi AI. Blood Pressure Goals in Acute Stroke-How Low Do You Go? Curr Hypertens Rep. 2018 Apr 10;20(4):28. doi: 10.1007/s11906-018-0827-5. PMID 29637385
- [Background] Gasecki D, Coca A, Cunha P, Hering D, Manios E, Lovic D, Zaninelli A, Sierra C, Kwarciany M, Narkiewicz K, Karaszewski B. Blood pressure in acute ischemic stroke: challenges in trial interpretation and clinical management: position of the ESH Working Group on Hypertension and the Brain. J Hypertens. 2018 Jun;36(6):1212-1221. doi: 10.1097/HJH.0000000000001704. PMID 29621070
- [Background] Jauch EC, Saver JL, Adams HP Jr, Bruno A, Connors JJ, Demaerschalk BM, Khatri P, McMullan PW Jr, Qureshi AI, Rosenfield K, Scott PA, Summers DR, Wang DZ, Wintermark M, Yonas H; American Heart Association Stroke Council; Council on Cardiovascular Nursing; Council on Peripheral Vascular Disease; Council on Clinical Cardiology. Guidelines for the early management of patients with acute ischemic stroke: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Mar;44(3):870-947. doi: 10.1161/STR.0b013e318284056a. Epub 2013 Jan 31. PMID 23370205
- [Derived] Georgianou E, Georgianos PI, Petidis K, Markakis K, Zografou I, Karagiannis A. Effect of Nebivolol and Olmesartan on 24-Hour Brachial and Aortic Blood Pressure in the Acute Stage of Ischemic Stroke. Int J Hypertens. 2019 Oct 7;2019:9830295. doi: 10.1155/2019/9830295. eCollection 2019. PMID 31687205